CLINICAL TRIAL: NCT00190606
Title: Efficacy and Safety of Duloxetine Compared With Placebo,Pelvic Floor Muscle Training, and Combined Duloxetine/Pelvic Floor Muscle Training in Subjects With Moderate to Sever Stress Urinary Incontinence
Brief Title: Efficacy and Safety of Duloxetine, Placebo and Pelvic Floor Muscle Training in Subjects With Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2615; F1J-MC-SBAF
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine
Procedure: Pelvic Floor Muscle Training (PFMT)
Procedure: Imitation PFMT
Drug: placebo

SUMMARY:
The study is a comparison of the efficacy and safety of duloxetine and pelvic floor muscle training with that of placebo in patients with moderate to severe stress urinary incontinence

ELIGIBILITY:
Inclusion Criteria:

* Female
* Between 18 and 75 years of age
* Confirmed pure genuine stress incontinence
* Have discrete episodes of incontinence
* Have pelvic organ prolapse of no greater than Stage II

Exclusion Criteria:

* Positive urine culture at visit 1
* Had formal PFMT with instruction
* Use of MAOI or other excluded medications
* Use of any anti-incontinence device, vaginal pessaries or any medication prescribed for the treatment of urinary incontinence

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2002-01; Study Completion 2006-04

PRIMARY OUTCOMES:
Effectiveness of combined duloxetine and PFMT with combined placebo and imitation PFMT in women with SUI as measured by percent change in Incontinence Episode Frequency from baseline to endpoint.
Effectiveness of combined duloxetine and PFMT with combined placebo and PFMT for up to 12 weeks in women with SUI as measured by percent change in Incontinence Episode Frequency from baseline to endpoint.

SECONDARY OUTCOMES:
Incontinence Quality of Life scores from baseline to endpoint.
Patient Global Impression - Impression at endpoint.
Symptoms Frequency & Bothersomeness.
Percent change in weekly continence pad usage (CPAD) from baseline to endpoint.
Change in Patient Satisfaction Questionnaires -2 and -4 questionnaire scores from baseline to endpoint.
Percent change in daily CPAD from baseline to endpoint.
Compare safety of duloxetine with placebo based on vital signs , laboratory values and the occurrence of treatment-emergent adverse events.
Compare combined duloxetine and PFMT, combined duloxetine and imitation PFMT, combined placebo with PFMT and combined placebo and imitation PFMTwith respect to efficacy and to safety.
Compare the effect of duloxetine and placebo on patient compliance to PFMT and imitation PFMT regimes using a daly patient-generated log of completed contractions.
Generate long-term safety data (during open-label extension) on duloxetine in the treatment of women with SUI.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Weston, Florida, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday - Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Nieuwegein, Netherlands